CLINICAL TRIAL: NCT01713244
Title: A Randomized Controlled Trial of Radiofrequency Ablation Assisted Hepatectomy and Hepatectomy Alone in the Treatment of Advanced Hepatocellular Carcinoma
Brief Title: Radiofrequency Ablation Assisted Hepatectomy Versus Hepatectomy Alone for Advanced Hepatocellular Carcinoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Southwest Hospital, China (Other)
Responsible Party: Principal Investigator, fengkai, Institute of Hepatobiliary Surgery, Southwest Hospital, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SKLKF201209
Record Dates: First submitted 2012-10-21; First posted 2012-10-24 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-11

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular Carcinoma; Radiofrequency Ablation; Hepatectomy; Recurrence
MeSH Terms: conditions — Carcinoma, Hepatocellular; Recurrence | interventions — Hepatectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hepatectomy (Active Comparator): Using Hepatectomy for the treatment of advanced HCC
  Interventions: Procedure: Hepatectomy
- RFA assisted Hepatectomy (Experimental): Ablating the liver tissue around the tumor before hepatectomy.
  Interventions: Procedure: RFA assisted Hepatectomy

INTERVENTIONS:
Procedure: RFA assisted Hepatectomy — Using RFA to ablate and block the small vessels around the tumor before resection to reduce the spreading of the cancer cell.
  Arms: RFA assisted Hepatectomy
Procedure: Hepatectomy — Treat the advanced HCC with the hepatectomy only.
  Arms: Hepatectomy

SUMMARY:
RFA has become a standard method in the treatment of small HCC(≤2 cm) due to its ease of use, safety, cost-effectiveness, and minimal invasiveness. It can ablated and blocked the small vessels while destroyed the tumor cell in situ. Surgical resection is the most widely accepted treatment for the patients with advanced hepatocellular carcinoma in the Asian countries. But the effectiveness of hepatectomy was depressed because of the high recurrence rate. The spreading of the cancer cell along the portal vein or the hepatic vein system during the operation account for the tumor recurrence. Using RFA to ablate and block the small vessels around the tumor before resection will reduce the spreading of the cancer cell. Investigators hypothesized that the RFA assisted hepatectomy might result in lower recurrence rate than hepatectomy alone in the treatment of advanced HCC. Thus, the purpose of this study was to prospectively compare the effects of RFA assisted hepatectomy with hepatectomy alone for the treatment of advanced HCC.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of HCC confirmed at our hospital.
2. Intrahepatic tumor count no higher than 3 and a minimum tumor diameter > 3 cm, but no more than 8cm.
3. Liver function of Child-Pugh Class A or B.
4. Tumors lacked intrahepatic and extrahepatic metastasis.
5. Tumors had not invaded the portal vein, the hepatic vein trunk or the secondary branches.
6. Indocyanine green retention at 15 minutes (ICG-15) of <10%.
7. No evidence of coagulopathy: platelet count > 50 × 109/L and a prolonged prothrombin time of < 5 seconds.
8. No other anti-tumor therapy received before the treatment. -

Exclusion Criteria:

1. Patients met the inclusion criteria but declined to participate.
2. Patients with severe portal hypertension, a history of esophageal variceal hemorrhage, severe hypersplenism syndrome, or refractory ascites.
3. Patients whose permanent pathology after treatment suggested metastatic liver cancer or primary liver cancer of another tissue type.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2012-10; Primary Completion 2016-10 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
Recurrence-free Survival | 2 years

SECONDARY OUTCOMES:
Overall Survival | 2 years

OTHER OUTCOMES:
Number of participants with adverse events | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Kuansheng Ma, Ph.D, Study Director — Institute of hepatobiliary surgery,Southwest Hospital
Locations (1):
- Institute of hepatobiliary surgery,Southwest Hospital, Chongqing, Chongqing Municipality, China